CLINICAL TRIAL: NCT02282436
Title: Muscle Atrophy in Patients With Chronic Obstructive Pulmonary DIsease : Substudy With Patients Who Experienced an Acute Exacerbation
Brief Title: Substudy : Patients With an Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Acronym: EXA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Annie Dubé, Professionnelle de recherche, Laval University
Other Study IDs: EXA-COPD-20765
Record Dates: First submitted 2014-10-09; First posted 2014-11-04 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood sample and muscle biopsy of vastus lateralis (quadriceps)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- COPD exacerbation: No specific intervention for this study
  Interventions: Other: No specific intervention for this study

INTERVENTIONS:
Other: No specific intervention for this study — No specific intervention for this study

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a leading cause of morbidity and mortality worldwide. Its prevalence is in progression and COPD is expected to become the fourth leading cause of death by 2030. COPD is characterized by periods of stability interspersed with acute infectious/inflammatory flare-ups, also called acute exacerbations, during which patients deteriorate, sometimes to the point of requiring immediate medical assistance. Although most patients eventually recover, repeated episodes of exacerbations may accelerate COPD progression. Exacerbations may further compromise the integrity of limb muscles by promoting further loss in muscle mass and strength.

The overall objective of this substudy is to elucidate how an acute COPD exacerbation may affect limb muscles.

DETAILED DESCRIPTION:
Focusing our attention during exacerbations, a period of aggravated systemic inflammation, should be more rewarding in terms of understanding the link between inflammation burst and muscle disease in COPD. We have recently acquired experimental data supporting a role for the ubiquitin proteasome pathway in the worsening of limb muscle structure and function during an acute exacerbation, providing a solid framework for this investigation. The overall objective of this proposal is to substantiate these preliminary findings and elucidate how systemic inflammation during acute COPD exacerbation may affect limb muscles. Ultimately, our research could open new therapeutic avenues to minimize the systemic consequences of an acute exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* COPD with an FEV1 of under 60% of predicted
* non-smoker
* between 50 and 75 years old
* experiencing an acute exacerbation of COPD (24-48 hours, before treatment)

Exclusion Criteria:

* all inflammatory disease (HIV, cancer, renal and cardiac deficiency)
* hormonal dysregulation
* inferior limb pathology
* neuromuscular pathology
* history of tobacco or alcool abuse
* oxygen dependent

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female who are experiencing an acute exacerbation of their COPD.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-05; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Increased levels of ubiquitin proteasome pathway proteins in patients experiencing an acute exacerbation of COPD | during an acute exacerbation of COPD (first 24-48 hours, before treatment)
  Our view is that targeting exacerbation is likely to unravel important mechanisms linking systemic inflammatory processes to downstream consequences on remote organs such as limb muscles. Inflammatory burst observed during exacerbation may be associated with upregulation of ubiquitin proteasome pathway (Atrogin-1, MuRF-1, Nedd4, ubiquitin C, poly-Ub), the main proteolytic pathway in this tissue, and thus with the occurrence of atrophying process.

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, PhD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Centre de recherche de l'Institut de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada